CLINICAL TRIAL: NCT03816917
Title: Discovery of Arthritis in Psoriasis Patients for Early Rheumatological Referral (DAPPER): a Cross-sectional Study
Brief Title: Discovery of Arthritis in Psoriasis Patients for Early Rheumatological Referral
Acronym: DAPPER
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Sint Maartenskliniek (Other)
Responsible Party: Sponsor
Other Study IDs: NL68137.091.18; Nederlands Trial Register (Registry Identifier: NTR7604)
Record Dates: First submitted 2018-12-27; First posted 2019-01-25 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2021-07

CONDITIONS: Psoriasis; Psoriatic Arthritis; Psoriasis Vulgaris; Psoriatic Nail
Keywords: Screening; Prediction Model
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic | interventions — Comorbidity; Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * serum
  * plasma
  * DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- topical treatment: 100 consecutive patients with cutaneous psoriasis, stratified on current therapy for cutaneous symptoms: only topical/UV therapy (no systemic therapy)
  Interventions: Other: cutaneous parameters of psoriasis (exposure); Other: comorbidity (exposure); Other: family history (exposure); Other: lifestyle (exposure); Other: patient reported outcomes (exposure); Other: inflammatory markers (exposure); Other: genetic (exposure)
- systemic treatment: 100 consecutive patients with cutaneous psoriasis, stratified on current therapy for cutaneous symptoms: systemic therapy, but no biologicals. Topical therapy is permitted.
  Interventions: Other: cutaneous parameters of psoriasis (exposure); Other: comorbidity (exposure); Other: family history (exposure); Other: lifestyle (exposure); Other: patient reported outcomes (exposure); Other: inflammatory markers (exposure); Other: genetic (exposure)
- biologics: 100 consecutive patients with cutaneous psoriasis, stratified on current therapy for cutaneous symptoms: systemic therapy with biologics. Other systemic and topical therapy is permitted.
  Interventions: Other: cutaneous parameters of psoriasis (exposure); Other: comorbidity (exposure); Other: family history (exposure); Other: lifestyle (exposure); Other: patient reported outcomes (exposure); Other: inflammatory markers (exposure); Other: genetic (exposure)

INTERVENTIONS:
Other: cutaneous parameters of psoriasis (exposure) — characteristic of the cutaneous domains of the psoriasis: age at start, disease duration, current and previous treatment PASI, BSA, nail involvement
Other: comorbidity (exposure) — medical and medication history, current and previous comorbidity
Other: family history (exposure) — Family history of PsC, PsA, IBD, AS, and uveitis
Other: lifestyle (exposure) — * Intoxications
  * Lifestyle: occupation and injuries, sport and physical hobbies
Other: patient reported outcomes (exposure) — VAS-score on fatigue, PsC severity, joint pain and general well-being
Other: inflammatory markers (exposure) — Measurements of inflammatory and bone remodeling markers in serum and plasma
Other: genetic (exposure) — Assessment of known HLA- and SNP-associations with PsA or PsA

SUMMARY:
Rationale: Psoriasis (PsO) is a common inflammatory skin disease. Besides the skin, it is recognized that this disease can affect multiple domains such as nails, joints and entheses. About 30% of the patients with PsO will develop symptoms in the musculoskeletal domains. Untreated inflammation in psoriatic arthritis (PsA) can lead to irreversible joint damage and further reduces quality of life. Since musculoskeletal involvement is often preceded by the dermatological symptoms of PsO, patients with pure cutaneous psoriasis (PsC) should be routinely screened for joint involvement. Current screening questionnaires, like the often used Psoriasis Epidemiology Screening Tool (PEST), offer a moderate discrimination between patients with PsA and PsC at best. Our aim is to assert the prevalence of known and previously undiagnosed PsA in a PsC cohort. By comparing the gathered data of the PsA and PsC patients, we hope to improve the screening of PsC patients, and to reduce both undertreatment of locomotor symptoms as well as unnecessary diagnostic investigations.

Objective: To ascertain the prevalence of PsA in a tertiary PsO cohort. Secondary objectives will be to ascertain the clinical features of these patients. With these features we want to find clinical, laboratory or genetic markers to predict the presence of PsA in PsO patients. Moreover, we wish to establish the added value of PsA screening for the quality of life (QoL) of PsO patients.

Study design: Multicenter cross-sectional study with a single follow-up visit after 1 year. Patients will be screened at baseline for PsA symptoms by a rheumatology resident and referred to a rheumatology clinic if deemed necessary. At baseline, several clinical and sociodemographic parameters will be assessed. We will collect blood samples for diverse biochemical studies and genomic DNA. Patients will be followed for 1 year after active screening for PsA. Quality of life (QoL) and treatment change will be recorded after this period, to assess the effect of screening and referral.

DETAILED DESCRIPTION:
This is a monocenter cohort study, which will span at least 1 year from inclusion to follow-up.

A sample of 300 patients known with PsC (cutaneous psoriasis) at the Department of Dermatology of the RadboudUMC, Nijmegen will be included. Inclusion of patients and collection of samples will be performed adjacent to their regular outpatient visits.

During screening, patients will be assessed for signs and symptoms of PsA (psoriatic arthritis). This will include a 68 tender joint count (TJC) and 66 swollen joint count (SJC), a dactylitis count, the Leeds enthesis index (LEI) and a questionnaire screening for inflammatory back pain (IBP).

At baseline visit, different parameters will be noted which can later be used to construct the prediction model. These will include sociodemographic data, relevant comorbidity, family history, characteristics of the PsC, intoxications, and constitutional and specific rheumatological signs and symptoms. During physical examination, the investigators will gather information about body measurements, skin and nail parameters, and rheumatological parameters.

Also, a screening questionnaires already in use (PEST) will be used, as well as a quality of life scores (PsAID12, DLQI, Short-Form 12 Health Survey/SF-12).

Blood will be drawn at baseline to check for different laboratory parameters which are associated with presence of PsA. Both inflammatory markers (e.g. cytokines, chemokines) as markers associated with bone metabolism are of interest. Also, DNA will be gathered via saliva and stored. At a later moment, this will be used to investigate the predictive value of different associated genetic polymorphisms and HLA-associations.

If there is a clinical suspicion of PsA in the clinical exam, the patient will be referred to the Department of Rheumatology of the Sint Maartenskliniek, Nijmegen (SMK). From there on, they will be included in PsA regular care. After 1 year, patient files of the referred patients will be checked to confirm the diagnosis. Also, treatment changes and their effect will be noted. This will include both clinical parameters of the PsA and QoL.

Patients already treated for PsA at a different clinic will not be referred to the SMK. They will be asked for permission to retrieve treatment-related data from their treating physician.

Patients without musculoskeletal involvement will be re-evaluated after 1 year. Again, treatment changes and quality of life will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cutaneous psoriasis
* Age 18 years or above
* Willing and able to comply with visits and study-related procedures
* Provide signed informed consent (IC)

Exclusion Criteria:

* Age below 18 years
* Unable to give IC
* Unable or unwilling to comply with visits and study-related procedures
* Participation in other trials involving PsO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cutaneous psoriasis, treated at a third line university outpatient dermatology clinic. Patients will be stratified based on current therapy.
Sampling Method: Non-Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
Presence of PsA according to CASPAR-criteria | at baseline
  The CASPAR-criteria are positive if a patient has inflammatory enthesitis OR peripheral OR axial arthritis AND cutaneous psoriasis (all of our patients) AND 1 additional outcome (see outcome 2 to 6)

SECONDARY OUTCOMES:
Presence of dactylitis | at baseline
  Dactylitis count, range 0-20, yes/no
Absence of rheumatoid factor | at baseline
  A rheumatoid factor measured in serum: U/mL, yes/no below the cutoff point as set by the local lab
Presence of new bone formation | at baseline
  X-rays of hand and feet as judged by the local radiologist, presence of new bone formation yes/no
Presence of typical psoriatic nail disease | at baseline
  NAPSI
Presence of typical psoriatic nail disease | at baseline
  N-NAIL
The presence of clinical enthesitis | at baseline
  Leeds Enthesitis Index, scored 0-6
The presence of arthritis | at baseline
  66 Swollen Joint Count, 0-66, yes/no
The presence of arthralgia | at baseline
  68 Tender Joint Count, 0-66, yes/no
The presence of inflammatory back pain | at baseline
  ASAS criteria for inflammatory back pain are positive is there is back pain for more than 3 months, and 4/5 of the following parameters are positive: age of onset <40 year, gradual development, improvement with exercise, no improvement with rest and back pain at night which improves on getting up

OTHER OUTCOMES:
Comorbidity | at baseline
  Score on Charlson Comorbidity Scale
Comorbidity | at baseline
  Score on Functional Comorbidity Index
Degree of cutaneous involvement | at baseline
  PASI
Degree of cutaneous involvement | at baseline
  Body surface (in percentage)
Quality of Life | at baseline and after 12 months
  Short Form 36 scores, DLQI scores, PsAID12 scores

CONTACTS AND LOCATIONS:
Overall Officials: Elke de Jong, Prof MD PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided